CLINICAL TRIAL: NCT03427411
Title: Phase II Trial of M7824 in Subjects With HPV Associated Malignancies
Brief Title: M7824 in Subjects With HPV Associated Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Julius Strauss, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180056; 18-C-0056
Record Dates: First submitted 2018-02-08; First posted 2018-02-09 (Actual); Results first posted 2022-02-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Human Papilloma Virus; Cervical Cancer; Oropharyngeal Cancer; Anal Cancer; Vaginal or Penile Cancer
Keywords: TGFR1 pathway signaling and overexpression; PD-1 inhibitors; Manageable Safety Profile; Bifunctional Fusion Protein; Refractory/Recurrent HPV Associated Malignancies
MeSH Terms: conditions — Uterine Cervical Neoplasms; Oropharyngeal Neoplasms; Anus Neoplasms; Penile Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Arm 1-M7824 1,200 mg intravenous (IV) once every 2 weeks (Experimental): M7824 at a flat dose of 1,200 mg intravenous (IV) once every 2 weeks
  Interventions: Drug: M7824

INTERVENTIONS:
Drug: M7824 — Flat dose of 1,200 mg of M7824 intravenous (IV) once every 2 weeks
  Other Names: MSB0011359C

SUMMARY:
Background:

In the United States, each year there are more than 30,000 cases of human papillomavirus (HPV) associated cancers. Some of these cancers are often incurable and are not improved by standard therapies. Researchers want to see if a new drug M7824, which targets and blocks a pathway that prevents the immune system from effectively fighting the cancer can shrink tumors in people with some HPV cancers.

Objectives:

To see if the drug M7824 causes tumors to shrink.

Eligibility:

Adults age 18 and older who have a cancer associated with HPV infection.

Design:

Participants will be screened with medical history and physical exam. They will review their symptoms and how they perform normal activities. They will have body scans. They will give blood and urine samples. They will have a sample of their tumor tissue taken if one is not available.

Participants will have an electrocardiogram to evaluate their heart. Then they will get the study drug through a thin tube in an arm vein.

Participants will get the drug every 2 weeks for 26 times (1 year). This is 1 course.

After the course, participants will be monitored but will not take the study drug. If their condition gets worse, they will start another course with the drug. This process can be repeated as many times as needed.

Treatment will stop if the participant has bad side effects or the drug stops working.

Throughout the study, participants will repeat some or all the screening tests.

After participants stop taking the drug, they will have a follow-up visit and repeat some screening tests. They will get periodic follow-up phone calls.

DETAILED DESCRIPTION:
Background:

* Metastatic or refractory/recurrent human papillomavirus (HPV) associated malignancies (cervical, anal, oropharyngeal cancers etc.) are often incurable and poorly palliated by standard therapies.

  * Transforming growth factor receptor type 1 (TGF R1) pathway signaling and overexpression are significantly associated with HPV+ cancers.
  * Programmed cell death protein 1 (PD-1) inhibitors have produced a 12-20% response rate for these diseases
  * M7824 is a novel bifunctional fusion protein composed of monoclonal antibodies against human programmed death-ligand 1 (PD- L1) and soluble extracellular domain of human TGF- receptor II (TGF- RII), which functions as a TGF- "trap."
  * Early data from a small cohort of patients with HPV associated malignancies in a phase I trial of M7824 has shown promising activity (NCT02517398). As of May 30, 2017, 4 of 9 patients (44%) with HPV associated malignancies have had preliminary evidence of clinical benefit including:
* Patient with metastatic cervical cancer with a 25% reduction in her disease at 3 months
* Patient with metastatic P16 positive (P16+) head and neck cancer with an unconfirmed partial response (PR) at 6 weeks
* Patient with metastatic anal cancer with a durable PR ongoing 9 months after starting treatment
* Patient with metastatic cervical cancer with a durable complete response (CR) ongoing 15 months after starting treatment.
* Notably, the P16+ head and neck cancer patient with unconfirmed PR, anal cancer patient with durable PR and cervical cancer patient with durable CR all have HPV+ disease.

  * Immune related adverse events with M7824 in the phase I trial to date have been on par with other PD-1/PD-L1 inhibitors, suggesting a manageable safety profile.
  * EMD Serono has an ongoing expansion cohort evaluating M7824 in patients with head and neck squamous cell carcinoma (HNSCC) as well as in cervical cancer excluding neuroendocrine cervical cancer.

Objective:

-To determine the objective response rate (ORR) according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) in subjects with recurrent or metastatic HPV associated malignancies.

Eligibility:

* Age greater than or equal to 18 years old
* Subjects with cytologically or histologically confirmed locally advanced or metastatic HPV

associated malignancies including:

* Non-Neuroendocrine Cervical cancers
* P16+ Oropharyngeal cancers
* Anal cancers
* Vulvar, vaginal, penile, squamous cell rectal and neuroendocrine cervical cancers
* Other locally advanced or metastatic solid tumors (e.g. lung, esophagus) that are known HPV+

  * Subjects must have measurable disease.

Design:

-This is a Phase II trial of M7824 in patients with recurrent or metastatic HPV associated

malignancies.

* Patients will be scheduled to receive 1,200 mg of M7824 intravenous (IV) every 2 weeks until off treatment criteria are met.
* There will be six cohorts: (1) Patients with anal cancer whose disease is naive to checkpoint inhibition, (2) Patients with non-neuroendocrine cervical cancer naive to checkpoint inhibition,

  (3) Patients with P16+ oropharyngeal cancers naive to checkpoint inhibition, and (4) Patients with other rare HPV associated tumors (e.g. squamous cell rectal, vulvar, vaginal, penile cancer, neuroendocrine cervical) naive to checkpoint inhibition, (5) Patients with any HPV associated cancers whose disease is refractory to checkpoint inhibition. Patients who are determined to be HPV negative after enrolling will be taken off of their previously assigned cohort and reassigned to cohort 6 and their slot on their previously assigned cohort will be replaced.
* Cohorts 1-5 of the trial will be conducted using a Simon two-stage phase II trial design.

ELIGIBILITY:
* INCLUSION CRITIERIA:
* Age greater than or equal to 18 years.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Subjects with cytologically or histologically confirmed locally advanced or metastatic human papillomavirus (HPV) associated malignancies including:

  * Non-Neuroendocrine Cervical cancers
  * P16 positive (P16+) Oropharyngeal cancers
  * Anal cancers
  * Vulvar, vaginal, penile, squamous cell rectal and neuroendocrine cervical cancers
  * Other locally advanced or metastatic solid tumors (e.g. lung, esophagus) that are known HPV+
* Patients must have disease that is not amenable to potentially curative resection
* Subjects must have measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Adequate hematologic function at screening, as follows:

  * Absolute neutrophil count (ANC) greater than or equal to 1 x 109/L
  * Hemoglobin greater than or equal to 9 g/dL
  * Platelets greater than or equal to 75,000/microliter.
* Adequate renal and hepatic function at screening, as follows:

  * Serum creatinine less than or equal to 1.5 x upper limit of normal (ULN) OR creatinine clearance (CrCl) greater than or equal to 40 mL/min per institutional standard
  * Bilirubin less than or equal to 1.5 x ULN OR in subjects with Gilbert's syndrome, a total bilirubin less than or equal to 3.0 x ULN
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 2.5 x ULN, unless liver metastases are present, then values must be less than or equal to 3 x ULN)
* The effects of M7824 on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and up to 60 days after the last dose of the drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Patients serologically positive for human immunodeficiency virus (HIV), Hep B, Hep C are eligible as long as the viral loads are undetectable by quantitative polymerase chain reaction (PCR). HIV positive patients must have cluster of differentiation 4 (CD4) count greater than or equal to 300 cells per cubic millimeter at enrollment, be on stable antiretroviral therapy and have no reported opportunistic infections within 12 months prior to enrollment.
* EXCLUSION CRITERIA:
* Pregnant women are excluded from this study because this drug has not been tested in pregnant women and there is potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to

treatment of the mother with M7824, breastfeeding should be discontinued if the mother is treated with M7824.

* Patients with prior investigational drug, chemotherapy, immunotherapy or any prior radiotherapy (except for palliative bone directed therapy) within the past 28 days prior to the first drug administration except if the investigator has assessed that all residual treatment-related toxicities have resolved or are minimal and feel the patient is otherwise suitable for enrollment. Patients may continue adjuvant hormonal therapy in the setting of a definitively treated cancer (e.g., breast).
* Major surgery within 28 days prior to the first drug administration (minimally invasive procedures such as diagnostic biopsies are permitted).
* Known intolerance to or life-threatening side effects resulting from prior checkpoint inhibitor therapy.
* Known active brain or central nervous system metastasis (less than 1 month out from definitive radiotherapy or surgery), seizures requiring anticonvulsant treatment (<3 months) or clinically significant cerebrovascular accident (<3 months). In order to be eligible patients must have repeat central nervous system (CNS) imaging at least two months after definitive treatment showing stable CNS disease. Patients with evidence of intra-tumoral or peritumoral hemorrhage on baseline imaging are also excluded unless the hemorrhage is grade less than or equal to 1 and has been shown to be stable on two consecutive imaging scans.
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent with exception of:

  * diabetes type I, eczema, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease or other mild autoimmune disorders not requiring immunosuppressive treatment;
  * Subjects requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses less than or equal to 10 mg of prednisone or equivalent per day;
  * Administration of steroids for other conditions through a route known to result in a minimal systemic exposure (topical, intranasal, intro-ocular, or inhalation) is acceptable;
  * Subjects on systemic intravenous or oral corticosteroid therapy with the exception of physiologic doses of corticosteroids (less than or equal to the equivalent of prednisone 10 mg/day) or other immunosuppressives such as azathioprine or cyclosporin A are excluded on the basis of potential immune suppression. For these subjects these excluded treatments must be discontinued at least 1 weeks prior to enrollment for recent short course use (less than or equal to 14 days) or discontinued at least 4 weeks prior to enrollment for long term use (>14 days). In addition, the use of corticosteroids as premedication for contrast enhanced studies is allowed prior to enrollment and on study.
* Subjects with a history of serious intercurrent chronic or acute illness, such as cardiac or pulmonary disease, hepatic disease, bleeding diathesis or recent (within 3 months) clinically significant bleeding events, or other illness considered by the Investigator as high risk for investigational drug treatment.
* History of non-HPV associated second malignancy within 3 years of enrollment except localized malignancy which has been adequately treated or malignancy which does not require active systemic treatment (e.g., low risk chronic lymphocytic leukemia (CLL).
* Known severe hypersensitivity reactions to monoclonal antibodies (Grade greater than or equal to 3 National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v4.03)
* Receipt of any organ transplantation requiring ongoing immunosuppression.
* Patients with vulvar cancer originating from differentiated vulvar intraepithelial neoplasia (d-VIN), as opposed to vulvar intraepithelial neoplasia of usual type, are excluded. Vulvar squamous cell carcinoma originating from differentiated VIN (d-VIN) is HPV negative; however, rare cases of HPV positive d-VIN can occur. Patients are not excluded if their tumor has tested positive for HPV or there is no documentation of prior VIN type.
* Patients with known HPV negative malignancies based on comprehensive laboratory testing (e.g. PCR based assay evaluating for HPV 16, 18, 31, 33, 35, 39, 51, 52, 56, 58, 59, 66, 68). Patients with HPV associated malignancies and unknown HPV status prior to enrollment are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julius Y Strauss, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP) .
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to the Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- [Background] Viens LJ, Henley SJ, Watson M, Markowitz LE, Thomas CC, Thompson TD, Razzaghi H, Saraiya M. Human Papillomavirus-Associated Cancers - United States, 2008-2012. MMWR Morb Mortal Wkly Rep. 2016 Jul 8;65(26):661-6. doi: 10.15585/mmwr.mm6526a1. PMID 27387669
- [Background] Levovitz C, Chen D, Ivansson E, Gyllensten U, Finnigan JP, Alshawish S, Zhang W, Schadt EE, Posner MR, Genden EM, Boffetta P, Sikora AG. TGFbeta receptor 1: an immune susceptibility gene in HPV-associated cancer. Cancer Res. 2014 Dec 1;74(23):6833-44. doi: 10.1158/0008-5472.CAN-14-0602-T. Epub 2014 Oct 1. PMID 25273091
- [Background] Wu P, Wu D, Li L, Chai Y, Huang J. PD-L1 and Survival in Solid Tumors: A Meta-Analysis. PLoS One. 2015 Jun 26;10(6):e0131403. doi: 10.1371/journal.pone.0131403. eCollection 2015. PMID 26114883
- [Derived] Strauss J, Gatti-Mays ME, Cho BC, Hill A, Salas S, McClay E, Redman JM, Sater HA, Donahue RN, Jochems C, Lamping E, Burmeister A, Marte JL, Cordes LM, Bilusic M, Karzai F, Ojalvo LS, Jehl G, Rolfe PA, Hinrichs CS, Madan RA, Schlom J, Gulley JL. Bintrafusp alfa, a bifunctional fusion protein targeting TGF-beta and PD-L1, in patients with human papillomavirus-associated malignancies. J Immunother Cancer. 2020 Dec;8(2):e001395. doi: 10.1136/jitc-2020-001395. PMID 33323462
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0056.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks: Participants with anal cancer, non-neuroendocrine cervical cancer, P16 positive (P16+) oropharyngeal cancers, and other rare HPV associated tumors (e.g., squamous cell rectal, vulvar, vaginal, penile cancer, neuroendocrine cervical) naïve to checkpoint inhibition treated with M7824 at a flat dose of 1,200 mg intravenous (IV) once every 2 weeks until confirmed progressive disease, death, unacceptable toxicity, or study withdrawal.
- Participants Refractory to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks: Participants with human papillomavirus (HPV) associated cancers refractory to checkpoint inhibition treated with M7824 at a flat dose of 1,200 mg intravenous (IV) once every 2 weeks until confirmed progressive disease, death, unacceptable toxicity, or study withdrawal.
Period: Overall Study
Arm/Group | Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks | Participants Refractory to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks
Started | 30 | 27
Completed | 30 | 26
Not Completed | 0 | 1
Not completed — Screen failure - platelets too low | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant enrolled in the refractory group was a screen failure and was not treated. However, collected baseline data is shown here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks | Participants Refractory to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks | Total
Number analyzed (Participants) | 30 | 27 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 18 | 43
  >=65 years | 5 | 9 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.48 (13.49) | 58.73 (11.94) | 55.96 (12.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 11 | 36
  Male | 5 | 16 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 28 | 25 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 23 | 26 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 30 | 27 | 57
Site of Primary Tumor [Count of Participants; unit: Participants]
  Anus | 4 | 6 | 10
  Cervix | 15 | 6 | 21
  Head-face or neck - Not Otherwise Specified | 1 | 1 | 2
  Head/Neck | 1 | 2 | 3
  Hypopharynx | 0 | 1 | 1
  Oropharynx | 0 | 1 | 1
  Rectum | 3 | 1 | 4
  Tongue | 0 | 1 | 1
  Tongue, Base of Tongue | 1 | 3 | 4
  Tonsil | 1 | 5 | 6
  Vagina | 1 | 0 | 1
  Vulva | 2 | 0 | 2
  Penile | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Achieved an Objective Confirmed Complete or Partial Overall Tumor Response
Description: The percentage of participants that achieved an objective confirmed complete or partial overall tumor response was measured using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Every six weeks for up to one year
Population: 1/30 participants was not evaluable in the naïve group because the participant was determined to be HPV negative. 1/27 was not evaluable in the refractory group because one participant was a screen failure and was not treated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks | Participants Refractory to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks
Number analyzed (Participants) | 29 | 26
percentage of participants | 31 [15.3 to 50.8] | 7.7 [0.9 to 25.1]

2. Secondary Outcome: Progression-free Survival Time (PFS)
Description: PFS is defined as the time from the date of first treatment to the date of disease progression or death. Progression was measured using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 and is defined as at least a 20% increase in the sum of diameters of target lesions, or appearance of one or more new lesions.
Time Frame: Time from the date of first treatment to the date of disease progression or death, up to 12 months
Population: 1/30 participants was not evaluable in the naïve group because they were found to be HPV negative and 1/27 was not evaluable in the refractory group because one participant was a screen failure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks | Participants Refractory to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks
Number analyzed (Participants) | 29 | 26
Months | 3.5 [1.5 to 7.4] | 1.4 [0.0 to 9.2]

3. Secondary Outcome: Percentage of Participants With Disease Control Who Achieved a Complete Response, Partial Response and Stable Disease Defined by the Response Evaluation Criteria in Solid Tumors (RECIST)Version 1.1 Lasting at Least 6 Months
Description: The percentage of participants with disease control who achieved a complete response, partial response and stable disease lasting at least 6 months was measured by the response evaluation criteria in solid tumors (RECIST)version 1.1. Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD) (at least a 20% increase in the sum of diameters of target lesions, or appearance of one or more new lesions).
Time Frame: 6 months
Population: 1/30 participants was not evaluable in the naïve group because they were determined to be HPV negative, and 1/27 was not evaluable in the refractory group because one participant was a screen failure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks | Participants Refractory to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks
Number analyzed (Participants) | 29 | 26
percentage of participants | 62.1 [42.3 to 79.3] | 19.2 [6.6 to 39.4]

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of first treatment to the date of death and was measured by Kaplan-Meier analysis.
Time Frame: Time from the date of first treatment to the date of death, up to 3 years.
Population: 1/30 participants was not evaluable in the naïve group because the patient was determined to be HPV negative, and 1/27 was not evaluable in the refractory group because one participant was a screen failure and was not treated.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks | Participants Refractory to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks
Number analyzed (Participants) | 29 | 26
Months | 19.2 [9.7 to NA] — The upper limit of the confidence interval cannot be estimated because several participants are still alive. | 4.4 [2.7 to 13.2]

5. Secondary Outcome: Number of Participants With Serious Grade ≥3 Adverse Events Considered Related to Study Treatment of M7824
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events version 5.0. A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 1 is mild. Grade 2 is moderate, Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: 28 days after treatment
Population: One participant enrolled in the refractory group was a screen failure and was not treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks | Participants Refractory to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks
Number analyzed (Participants) | 30 | 26
Participants | 6 | 4

6. Secondary Outcome: Number of Checkpoint Inhibitor Naive Participants With Response Based on Adequate Similarity (Defined as P-value > 0.2 With Fisher's Exact Test) of Results in Cohorts 1 and 2
Description: Response based on adequate similarity defined as P-value > 0.2 with Fisher's exact test of results in cohorts 1 and 2 was compared with a two-sided Fishers exact test, and response was measured by the response evaluation criteria in solid tumors (RECIST)version 1.1. Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease is at least a 20% increase in the sum of diameters of target lesions, or appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD).
Time Frame: median of 2 years
Population: Only cohorts 1 and 2 was evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks
Number analyzed (Participants) | 29
Participants
  Complete Response | 2
  Partial Response | 7
  Progressive Disease | 10
  Stable Disease | 9
  Not Evaluable | 1
Statistical Analysis 1: Comparison: Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks; Test type: Non-Inferiority — Non-inferiority was defined as response rates which were sufficiently similar (p>0.20 by Fisher's exact test); p = 0.6143, Fisher Exact — The p value was calculated and was 0.6143 which is > 0.2 (pre-defined threshold)

7. Secondary Outcome: Percentage of Participants That Were Hospitalized Because of Adverse Events Attributed to Disease Progression
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Disease progression is at least a 20% increase in the sum of diameters of target lesions, or appearance of one or more new lesions measured by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: Up to 30 days from last treatment
Population: One participant enrolled in the refractory group was a screen failure and was not treated.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks | Participants Refractory to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks
Number analyzed (Participants) | 30 | 26
percentage of participants | 37.9 | 69.2

8. Secondary Outcome: Duration of Response (Complete Response or Partial Response)
Description: Duration of response is defined as the time from complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease (PD) is objectively documented. Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progression is at least a 20% increase in the sum of diameters of target lesions, or appearance of one or more new lesions.
Time Frame: Time from complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease (PD) is objectively documented, up to 12 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks | Participants Refractory to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks
Number analyzed (Participants) | 9 | 2
Months | NA [8.3 to NA] — Median and upper end of the confidence interval cannot be estimated because duration of response was censored at the time of data cut off in 6/9 responders since these 6 participants have not had disease recurrence and therefore did not have a duration of response. The other 20 participants on this cohort were not assessed for duration of response as they did not have a response to begin with. Therefore median duration of response and upper end of the confidence interval cannot be calculated. | 4.0 [2.8 to NA] — The upper end of the confidence interval cannot be estimated because of the low number of responding participants (n=2) assessed for duration of response in this cohort. In addition, the other 24 participants on this cohort were not assessed for duration of response as they did not have a response to begin with. Therefore the upper end of the confidence interval cannot be calculated.

9. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 42 months and 28 days for the naïve group, and 40 months and 16 days for the refractory group.
Population: One enrolled participant was a screen failure and was not treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks | Participants Refractory to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks
Number analyzed (Participants) | 30 | 26
Participants | 30 | 26

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 42 months and 28 days for the naïve group, and 40 months and 16 days for the refractory group.
Description: One participant enrolled in the refractory group was a screen failure and was not treated.
Arm/Group | Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks | Participants Refractory to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks
All-Cause Mortality (participants affected / at risk) | 18/30 | 22/26
Serious Adverse Events (participants affected / at risk) | 19/30 | 21/26
Other Adverse Events (participants affected / at risk) | 30/30 | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks (N=30) | Participants Refractory to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks (N=26)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 3 (5)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (6) | 6 (12)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Death Not Otherwise Specified (NOS) (General disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 0 (0) | 5 (5)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 3 (4)
Fever (General disorders) | 1 (1) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fungemia (Infections and infestations) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Hepatobiliary disorders - Other, Hepatic duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, Nodular Regenerative Hyperplasia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, left hepatic lobe abscesses (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 1 (2) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Death due to disease progression reported to principal investigator on 8/16/18
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) — Neoplasm, Malignant, Metastatic Rectal Cancer
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, brain metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — disease progression head and neck squamous cell carcinoma (HNSCC)
Nervous system disorders - Other, Vocal fold paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, balance difficulties (Nervous system disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, Specify (Renal and urinary disorders) | 0 (0) | 1 (1) — Hydronephrosis secondary to UT obstruction-stent replacement indicated
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 1 (1)
Surgical and medical procedures - Other, Left Psoas Mass Resection (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Nephrostomy tube exchange trauma (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Resection abdominal (abd) wall mets (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Resection abd wall mets w/abd wall reconstruction (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, TAVR aortic valve replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, craniotomy for resection of cerebellar tumors (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, radiation therapy for cerebellar tumor (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, surgery to stabilize leg bone metastasis (Surgical and medical procedures) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Naïve to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks (N=30) | Participants Refractory to Checkpoint Inhibition - M7824 1,200 mg Intravenous Once Every 2 Weeks (N=26)
Abdominal pain (Gastrointestinal disorders) | 8 (11) | 7 (10)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (5) | 4 (4)
Alkaline phosphatase increased (Investigations) | 1 (1) | 4 (4)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 19 (44) | 19 (53)
Anorexia (Metabolism and nutrition disorders) | 10 (10) | 12 (16)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (2)
Ascites (Gastrointestinal disorders) | 3 (5) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (8) | 4 (6)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (10) | 4 (4)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (3) | 1 (1)
Blurred vision (Eye disorders) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 2 (2) | 1 (3)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
CPK increased (Investigations) | 1 (3) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Chills (General disorders) | 2 (3) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Concentration impairment (Nervous system disorders) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 4 (6)
Constipation (Gastrointestinal disorders) | 10 (11) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 5 (8)
Creatinine increased (Investigations) | 3 (3) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (4) | 7 (8)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (16) | 4 (5)
Dizziness (Nervous system disorders) | 4 (4) | 5 (6)
Dry eye (Eye disorders) | 1 (4) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (3) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 3 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 11 (14)
Ear and labyrinth disorders - Other, Continuous drainage L ear; hospitalized (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, Intermittent bloody discharge L ear (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, Specify (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Intermittent serous and sanguineous discharge L ear s/p Myringotomy; Ofloxacin indicated
Ear and labyrinth disorders - Other, Left ear fullness/congestion-ENT consult ordered (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, fullness/congestion left ear (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 8 (9) | 3 (4)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 4 (4)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Extrapyramidal disorder (Nervous system disorders) | 2 (2) | 0 (0)
Eye disorders - Other, peripheral visual fields altered left eye, r/t brain lesion (Eye disorders) | 1 (1) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 3 (4)
Fatigue (General disorders) | 18 (32) | 11 (14)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 7 (11) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Flashing lights (Eye disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (2)
Flu like symptoms (General disorders) | 6 (7) | 3 (3)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
Gait disturbance (General disorders) | 2 (2) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other, Diverticulosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Esophageal erosions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, Hyperpigmentation of tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 9 (10) | 4 (4)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 5 (8) | 3 (3)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 5 (6) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (4)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (9) | 8 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 7 (14) | 3 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (4) | 3 (5)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 6 (12)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 6 (11)
Hypotension (Vascular disorders) | 0 (0) | 4 (4)
Hypothyroidism (Endocrine disorders) | 7 (8) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 1 (1)
Infections and infestations - Other, Specify (Infections and infestations) | 1 (1) | 0 (0) — Diagnosed with Influenza A associated with malaise, nausea and interim fever; Tamiflu indicated
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (5)
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (3) | 1 (2)
Lung infection (Infections and infestations) | 1 (1) | 1 (2)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 11 (22) | 12 (27)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (6) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, TMJ symptoms, Left jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, partial tendon rupture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 11 (18) | 8 (10)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Benign Keratoacanthomas back of neck and R clavicle-dermatology (DERM) consult and monitoring
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Brain lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Dermal carcinoma with lymphovascular invasion (LVI) on forehead, mid-back, and abdomen (R lateral and superior chest)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — KERATOACANTHOMA, right forearm
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Keratoacanthoma lesions as per Dermatology bx results; steroid cream and prednisone indicated
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Keratoacanthoma on face & neck
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Keratoacanthoma on face/neck-cryotherapy indicated on 11/6/18
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Keratoacanthoma, site left upper eyelid
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Keratoacanthomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Keratoacanthomas (left shoulder)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Keratoacanthomas, bilateral arms, chest, back, neck per Derm dx; study drug held beg 10/23/18
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Keratoacanthomas; liquid nitrogen to lesions on nose, R knee; neck +R chest lesions resolved
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Per DERM, described as clinically a Keratoacanthoma
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nervous system disorders - Other, Specify (Nervous system disorders) | 1 (1) | 0 (0) — Withdrawal sys: tremulousness, fever, chills since stoppage of MS Contin
Nervous system disorders - Other, balance difficulties (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (16) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Oral hemorrhage (Gastrointestinal disorders) | 9 (10) | 6 (9)
Oral pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 6 (9) | 3 (3)
Pain in extremity (General disorders) | 3 (7) | 6 (7)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 2 (3)
Pelvic pain (Reproductive system and breast disorders) | 2 (5) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Perineal pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (14) | 8 (16)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 10 (17) | 6 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (16) | 1 (1)
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 6 (11) | 3 (3)
Rectal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Renal and urinary disorders - Other, Specify (Renal and urinary disorders) | 1 (1) | 0 (0) — Bacteriuria as per urine culture collected per Urology Consult; negative for infection
Renal and urinary disorders - Other, Hydronephrosis-moderate, L-sided (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, Urinary hesitancy and sensation of incomplete voiding (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Intermittent hemoptysis; Lovenox dose adjustment indicated-Low-molecular-weight heparin (LMWH) dose initiated
Respiratory, thoracic and mediastinal disorders - Other, Specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Intermittent sneezing and rhinorrhea which resolve with Tylenol
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 1 (2) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 7 (7)
Skin and subcutaneous tissue disorders - Other, seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 3 (3) | 1 (1)
Skin papilloma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, inguinal hernia (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, surgical de-bulking condyloma (Surgical and medical procedures) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 4 (5) | 6 (6)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (3) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 3 (5) | 2 (2)
Vision decreased (Eye disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (12) | 8 (11)
Weight gain (Investigations) | 2 (7) | 1 (1)
Weight loss (Investigations) | 6 (14) | 7 (10)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 3 (4) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT03427411/Prot_SAP_000.pdf
  • Informed Consent Form: Screening Consent (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT03427411/ICF_001.pdf
  • Informed Consent Form: Affected Patient Consent (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT03427411/ICF_002.pdf